CLINICAL TRIAL: NCT06144827
Title: Pilot Study to Assess the Role of Blood-based Biomarkers and Quantitative MR Imaging for Patients Receiving Radiation Therapy for Liver Cancer
Brief Title: A Pilot Study For Patients Receiving Radiation Therapy for Liver Cancer
Acronym: HepQuant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI indicated that the site was unable to procure shunt. No participants were enrolled and this HepQuant study will be withdrawn.
Sponsor: Montefiore Medical Center (Other)
Collaborators: HepQuant, LLC (Industry); Perspectum (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-14687
Record Dates: First submitted 2023-11-08; First posted 2023-11-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cancer, Hepatocellular; Radiotherapy Side Effect
MeSH Terms: conditions — Liver Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Multiparametric MRI scan group (Active Comparator): Multiparametric MRI scans will be used to evaluate baseline degree of liver fibroinflammation and function as well as temporal changes in liver fibroinflammation and function using MRI-based LiverMultiScan software.
  Interventions: Device: Multiparametric MRI scans
- Multiparametric MRI scans + HepQuantShunt Test group (Experimental): Eligible patients can have previously undergone any modality and number of prior treatments for their hepatic malignancies, must be considered for either liver photon or proton radiation in the de-novo or re-irradiation setting and can be simultaneously enrolled on parallel trials.
  Interventions: Device: Multiparametric MRI scans; Device: Multiparametric MRI scans + HepQuantShunt Test

INTERVENTIONS:
Device: Multiparametric MRI scans — Multiparametric MRI scans will be used to evaluate baseline degree of liver fibroinflammation and function as well as temporal changes in liver fibroinflammation and function using MRI-based LiverMultiScan software. We will also measure liver function using HepQuant SHUNT test in a subset of patients enrolled in this study.
Device: Multiparametric MRI scans + HepQuantShunt Test — Eligible patients can have previously undergone any modality and number of prior treatments for their hepatic malignancies, must be considered for either liver photon or proton radiation in the de-novo or re-irradiation setting and can be simultaneously enrolled on parallel trials. Patients must not have any contraindications that would preclude MRI imaging or receipt of HepQuant SHUNT test for those agreeable to have HepQuant SHUNT test.
  Arms: Multiparametric MRI scans + HepQuantShunt Test group

SUMMARY:
The purpose of this study is to evaluate the role of quantitative MR imaging and blood-based biomarkers to measure liver function in patients receiving radiation therapy for liver cancer or cancer that has spread to the liver.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the role of quantitative MR imaging and blood-based biomarkers to measure liver function in patients receiving radiation therapy for liver cancer or cancer that has spread to the liver. The feasibility of using MR imaging to monitor liver function at baseline and following liver radiation therapy will be determined. Information from MR images and blood samples, along with patient questionnaires, will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patient has the psychological ability and general health needed to provide informed consent, completion of study requirements, and required follow-up
* Patient provides study-specific informed consent prior to study entry
* All primary histologies (Hepatocellular carcinoma or Cholangiocarcinoma) as well as hepatic metastases are eligible
* Prior history of radiation therapy (external beam or radioembolization) is allowed, with no limit to the number of prior courses of radiation therapy
* Any number of lesions (with no size limit) of pathologically documented (histologically or cytologically) or radiographically proven tumor/metastasis that are being targeted
* Prior history of chemotherapy, immunotherapy, or targeted biological therapy is allowed
* Concurrent enrollment on other prospective registry or treatment intention trials is allowed

Exclusion Criteria:

* Pregnant or breast-feeding females
* Subjects with history of claustrophobia impacting ability to perform MRI during the study
* Subjects who fulfill any of the contraindications for MRI; examples include any ferromagnetic material, any metallic shrapnel or fragments or implanted electronic devices contained within the body or metal-containing tattoos
* Unable to participate in MR assessments due to physical limitations of equipment tolerances (MRI bore size and/or weight limit)
* Any person unable to lie still within the environment of the MRI scanner or maintain a breath hold for the required period to acquire images

Exclusion criteria for HepQuant SHUNT testing ONLY:

* Known history or suspected hypersensitivity to human serum albumin, or its preparations
* Subjects with extensive resection of large segments of small intestine (short gut) or severe gastroparesis
* Subjects on either a non-selective beta blocker (propranolol, nadolol) or an angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) who are unwilling or unable to delay taking their normal dose the morning of their testing
* Subjects who are allergic to any ingredient in the formulations or components in the HepQuant SHUNT kit including human serum albumin (HSA) or cholate compounds (theoretical - none yet reported)
* Subjects unwilling or unable to fast for at least 5 hours. Fasting means no intake of food or food supplements, including fiber preparations or biosimilars; or, any preparations or resins (cholestyramine, colestipol, colesalvalem) that might act within the gut lumen to bind the orally administered d4-cholate in the HepQuant test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Quantitative Multiparametric MRI | Up to 12 Months
  Feasibility will be determined by assessing the percentage of patients who complete at least two quantitative multiparametric MRI scans after study enrollment. The feasibility endpoint will be presented as proportions and a Clopper Pearson 95% exact confidence interval will be determined.

SECONDARY OUTCOMES:
Change in Disease Severity Index (DSI) scores | Baseline and 3 months post-RT
  Change in DSI scores from baseline will be evaluated using HepQuant SHUNT testing. The HepQuant SHUNT test measures hepatocyte function using the Disease Severity Index (DSI). Increased DSI scores have been correlated with worsening liver function and disease severity and progression and response to treatments. The DSI calculation is proprietary; however, the test generates a liver DSI score ranging from 0 (no hepatic impairment) to 50 (severe hepatic impairment) that is a composite of both hepatic filtration rates and correlates with stage of fibrosis, presence of varices, and risk for future clinical outcomes. Raw changes in DSI scoring from baseline scores will be summarized using descriptive statistics and will be examined using a paired t-test or Wilcoxon Sign rank test.
Ability of LiverMultiScan™ MRI software to predict the risk of non-classic radiation-induced liver disease (RILD) by measuring the pre-RT liver health assessment score | Baseline to 6 Months post-RT
  The ability of LiverMultiScan to predict the risk of non-classic RILD will be evaluated. The pre-radiotherapy liver health assessment score will be calculated by measuring the Future Liver Remnant volume outside the 50% radiation isodose line weighted by the liver cT1 value. MRI images will be post-processed using LiverMultiScan, which provides a multiparametric quantitative map of a region of interest in the liver including characterization of the underlying liver fibroinflammation as reported by a corrected T1 (cT1) value, which will be measured and reported in milliseconds (ms). The likelihood of non-classic RILD based on the cT1 value will be assessed using multivariable logistic regression.
  Non-classic RILD is defined as either worsening of Child-Pugh Score by >=2 points (overall range: 5-15 points) at 6 months following RT or an elevated aminotransferase (ALT or AST) level > 5 times the upper limit of normal or baseline value within 90 days of completion of RT.
Change in Total Liver Volume and Volume of non-irradiated and irradiated lobes | Baseline and 3, 6, 9, and 12 Months post-RT
  Change in total liver volume, as well as volume of non-irradiated and irradiated liver lobes, from pre-radiotherapy treatment at baseline will be evaluated using Gd-EOB-DTPA enhanced MRI of the abdomen at the specified timeframes to assess the impact of radiotherapy. Mean changes in total liver volume (cm^3) and volume of non-irradiated and irradiate lobes will be assessed using the MRI software image analysis and summarized by study arm. The data will be analyzed using linear mixed-effects models. Increases in liver volume are correlated to more favorable outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Rafi Kabbarriti, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Russell AH, Clyde C, Wasserman TH, Turner SS, Rotman M. Accelerated hyperfractionated hepatic irradiation in the management of patients with liver metastases: results of the RTOG dose escalating protocol. Int J Radiat Oncol Biol Phys. 1993 Sep 1;27(1):117-23. doi: 10.1016/0360-3016(93)90428-x. PMID 8365932
- [Background] Ben-Josef E, Lawrence TS. Radiotherapy for unresectable hepatic malignancies. Semin Radiat Oncol. 2005 Oct;15(4):273-8. doi: 10.1016/j.semradonc.2005.04.006. PMID 16183481
- [Background] Dawson LA, Guha C. Hepatocellular carcinoma: radiation therapy. Cancer J. 2008 Mar-Apr;14(2):111-6. doi: 10.1097/PPO.0b013e31816a0e80. PMID 18391616
- [Background] Ohri N, Tome WA, Mendez Romero A, Miften M, Ten Haken RK, Dawson LA, Grimm J, Yorke E, Jackson A. Local Control After Stereotactic Body Radiation Therapy for Liver Tumors. Int J Radiat Oncol Biol Phys. 2021 May 1;110(1):188-195. doi: 10.1016/j.ijrobp.2017.12.288. Epub 2018 Jan 6. PMID 29395629
- [Background] Tse RV, Hawkins M, Lockwood G, Kim JJ, Cummings B, Knox J, Sherman M, Dawson LA. Phase I study of individualized stereotactic body radiotherapy for hepatocellular carcinoma and intrahepatic cholangiocarcinoma. J Clin Oncol. 2008 Feb 1;26(4):657-64. doi: 10.1200/JCO.2007.14.3529. Epub 2008 Jan 2. PMID 18172187
- [Background] Miften M, Vinogradskiy Y, Moiseenko V, Grimm J, Yorke E, Jackson A, Tome WA, Ten Haken RK, Ohri N, Mendez Romero A, Goodman KA, Marks LB, Kavanagh B, Dawson LA. Radiation Dose-Volume Effects for Liver SBRT. Int J Radiat Oncol Biol Phys. 2021 May 1;110(1):196-205. doi: 10.1016/j.ijrobp.2017.12.290. Epub 2018 Jan 6. PMID 29482870
- [Background] Bujold A, Massey CA, Kim JJ, Brierley J, Cho C, Wong RK, Dinniwell RE, Kassam Z, Ringash J, Cummings B, Sykes J, Sherman M, Knox JJ, Dawson LA. Sequential phase I and II trials of stereotactic body radiotherapy for locally advanced hepatocellular carcinoma. J Clin Oncol. 2013 May 1;31(13):1631-9. doi: 10.1200/JCO.2012.44.1659. Epub 2013 Apr 1. PMID 23547075
- [Background] Andolino DL, Johnson CS, Maluccio M, Kwo P, Tector AJ, Zook J, Johnstone PA, Cardenes HR. Stereotactic body radiotherapy for primary hepatocellular carcinoma. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e447-53. doi: 10.1016/j.ijrobp.2011.04.011. Epub 2011 Jun 7. PMID 21645977
- [Background] Su TS, Luo R, Liang P, Cheng T, Zhou Y, Huang Y. A prospective cohort study of hepatic toxicity after stereotactic body radiation therapy for hepatocellular carcinoma. Radiother Oncol. 2018 Oct;129(1):136-142. doi: 10.1016/j.radonc.2018.02.031. Epub 2018 Mar 13. PMID 29548558
- [Background] Hasan S, Thai N, Uemura T, Kudithipudi V, Renz P, Abel S, Kirichenko AV. Hepatocellular carcinoma with child Pugh-A Cirrhosis treated with stereotactic body radiotherapy. World J Gastrointest Surg. 2017 Dec 27;9(12):256-263. doi: 10.4240/wjgs.v9.i12.256. PMID 29359031
- [Background] Nabavizadeh N, Waller JG, Fain R 3rd, Chen Y, Degnin CR, Elliott DA, Mullins BT, Patel IA, Dyer BA, Fakhoury K, Naugler WE, Farsad K, Tanyi JA, Fuss M, Thomas CR Jr, Hung AY. Safety and Efficacy of Accelerated Hypofractionation and Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma Patients With Varying Degrees of Hepatic Impairment. Int J Radiat Oncol Biol Phys. 2018 Mar 1;100(3):577-585. doi: 10.1016/j.ijrobp.2017.11.030. Epub 2017 Nov 27. PMID 29413273
- [Background] Cheng JC, Wu JK, Huang CM, Huang DY, Cheng SH, Lin YM, Jian JJ, Yang PS, Chuang VP, Huang AT. Radiation-induced liver disease after radiotherapy for hepatocellular carcinoma: clinical manifestation and dosimetric description. Radiother Oncol. 2002 Apr;63(1):41-5. doi: 10.1016/s0167-8140(02)00061-0. PMID 12065102
- [Background] Hollebecque A, Cattan S, Romano O, Sergent G, Mourad A, Louvet A, Dharancy S, Boleslawski E, Truant S, Pruvot FR, Hebbar M, Ernst O, Mathurin P. Safety and efficacy of sorafenib in hepatocellular carcinoma: the impact of the Child-Pugh score. Aliment Pharmacol Ther. 2011 Nov;34(10):1193-201. doi: 10.1111/j.1365-2036.2011.04860.x. Epub 2011 Sep 29. PMID 21958438
- [Background] Cardenes HR, Price TR, Perkins SM, Maluccio M, Kwo P, Breen TE, Henderson MA, Schefter TE, Tudor K, Deluca J, Johnstone PA. Phase I feasibility trial of stereotactic body radiation therapy for primary hepatocellular carcinoma. Clin Transl Oncol. 2010 Mar;12(3):218-25. doi: 10.1007/s12094-010-0492-x. PMID 20231127
- [Background] Culleton S, Jiang H, Haddad CR, Kim J, Brierley J, Brade A, Ringash J, Dawson LA. Outcomes following definitive stereotactic body radiotherapy for patients with Child-Pugh B or C hepatocellular carcinoma. Radiother Oncol. 2014 Jun;111(3):412-7. doi: 10.1016/j.radonc.2014.05.002. Epub 2014 Jun 3. PMID 24906626
- [Background] Weiner AA, Olsen J, Ma D, Dyk P, DeWees T, Myerson RJ, Parikh P. Stereotactic body radiotherapy for primary hepatic malignancies - Report of a phase I/II institutional study. Radiother Oncol. 2016 Oct;121(1):79-85. doi: 10.1016/j.radonc.2016.07.020. Epub 2016 Aug 23. PMID 27566894
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Pavlides M, Banerjee R, Sellwood J, Kelly CJ, Robson MD, Booth JC, Collier J, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging predicts clinical outcomes in patients with chronic liver disease. J Hepatol. 2016 Feb;64(2):308-315. doi: 10.1016/j.jhep.2015.10.009. Epub 2015 Nov 10. PMID 26471505
- [Background] Jayaswal ANA, Levick C, Collier J, Tunnicliffe EM, Kelly MD, Neubauer S, Barnes E, Pavlides M. Liver cT1 decreases following direct-acting antiviral therapy in patients with chronic hepatitis C virus. Abdom Radiol (NY). 2021 May;46(5):1947-1957. doi: 10.1007/s00261-020-02860-5. Epub 2020 Nov 28. PMID 33247768
- [Background] Janowski K, Shumbayawonda E, Dennis A, Kelly M, Bachtiar V, DeBrota D, Langford C, Thomaides-Brears H, Pronicki M, Grajkowska W, Wozniak M, Pawliszak P, Chelstowska S, Jurkiewicz E, Banerjee R, Socha P. Multiparametric MRI as a Noninvasive Monitoring Tool for Children With Autoimmune Hepatitis. J Pediatr Gastroenterol Nutr. 2021 Jan 1;72(1):108-114. doi: 10.1097/MPG.0000000000002930. PMID 32925554
- [Background] Mole DJ, Fallowfield JA, Sherif AE, Kendall T, Semple S, Kelly M, Ridgway G, Connell JJ, McGonigle J, Banerjee R, Brady JM, Zheng X, Hughes M, Neyton L, McClintock J, Tucker G, Nailon H, Patel D, Wackett A, Steven M, Welsh F, Rees M; HepaT1ca Study Group. Quantitative magnetic resonance imaging predicts individual future liver performance after liver resection for cancer. PLoS One. 2020 Dec 2;15(12):e0238568. doi: 10.1371/journal.pone.0238568. eCollection 2020. PMID 33264327
- [Background] Sethi P, Thavanesan N, Welsh FK, Connell J, Pickles E, Kelly M, Fallowfield JA, Kendall TJ, Mole DJ, Rees M. Quantitative multiparametric MRI allows safe surgical planning in patients undergoing liver resection for colorectal liver metastases: report of two patients. BJR Case Rep. 2021 Jan 12;7(3):20200172. doi: 10.1259/bjrcr.20200172. eCollection 2021 May 1. PMID 34131498
- [Background] Everson GT, Shiffman ML, Hoefs JC, Morgan TR, Sterling RK, Wagner DA, Lauriski S, Curto TM, Stoddard A, Wright EC; HALT-C Trial Group. Quantitative liver function tests improve the prediction of clinical outcomes in chronic hepatitis C: results from the Hepatitis C Antiviral Long-term Treatment Against Cirrhosis Trial. Hepatology. 2012 Apr;55(4):1019-29. doi: 10.1002/hep.24752. Epub 2012 Mar 1. PMID 22030902
- [Background] Burton JR Jr, Helmke S, Lauriski S, Kittelson J, Everson GT. The within-individual reproducibility of the disease severity index from the HepQuant SHUNT test of liver function and physiology. Transl Res. 2021 Jul;233:5-15. doi: 10.1016/j.trsl.2020.12.010. Epub 2021 Jan 2. PMID 33400995